CLINICAL TRIAL: NCT04355637
Title: Treatment With Inhaled Corticosteroids in Patients Hospitalized Because of COVID19 Pneumonia
Brief Title: Inhaled Corticosteroid Treatment of COVID19 Patients With Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sara Varea (Other)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACTIC-COVID; 2020-001616-18 (EudraCT Number)
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): patients receiving standard of care to treat their pneumonia
- Intervention (Experimental): patients receiving standard of care to treat their pneumonia + inhaled budesonide
  Interventions: Drug: Inhaled budesonide

INTERVENTIONS:
Drug: Inhaled budesonide — adding budesonide to standard of care for pneumonia in COVID19 positive patients
  Arms: Intervention

SUMMARY:
Randomized, prospective, controlled open label clinical trial aimed at investigating if the addition of inhaled corticosteroids (budesonide) reduces treatment failure (defined as a composite variable by the initiation of treatment with high flow-O2 therapy, non-invasive or invasive ventilation, systemic steroids, use of biologics (anti IL-6 or anti IL-1) and/or death) according to hospital standard of care guidance) at day 15 after initiation of therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* COVID19 positive
* hospitalized because of pneumonia (status #3 - #4 World Health Organization (WHO) scale)
* without contraindications to receive study treatment
* informed consent

Exclusion Criteria:

* receiving corticoids (inhaled or systemic)
* receiving anti Interleukin-1 (IL-1) or anti-IL-6 drugs
* receiving high flow oxygen therapy
* receiving mechanical ventilation
* pregnancy
* participating in another intervention trial for COVID19

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in both arms fulfilling the criteria for treatment failure | 15 days after treatment
  composite variable that includes the initiation of treatment with high flow-O2 therapy, non-invasive or invasive ventilation and/or death) at day 15 after initiation of therapeutic intervention

SECONDARY OUTCOMES:
ICU admission | baseline, day 3, day 7, day 15, day 30
  Yes/no
ICU refusal | baseline, day3, day 7, day 15, day 30
  yes/no and reason
Occurrence of complications | baseline, day3, day 7, day 15, day 30
  infectious cardiovascular and /or metabolic complications as well as variation in the 7 point WHO scale.
lactate dehydrogenase (LDH) | at baseline, day 3, day 7, day 15, day 30
  U/L
C Reactive Protein (CRP) | at baseline, day 3, day 7, day 15, day 30
  mg/dL
ferritin | at baseline, day 3, day 7, day 15, day 30
  ng/mL
D-dimer | at baseline, day 3, day 7, day 15, day 30
  ng/mL
leukocyte counts | at baseline, day 3, day 7, day 15, day 30
  x10^9/L

CONTACTS AND LOCATIONS:
Locations (14):
- Argentina (7):
  - Hospital de Infecciosas "Francisco Javier Muñiz", Ciudad Autonoma de Buenos Aires, Buenos Aires
  - CEMIC (Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno"), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital de Rehabilitación Respiratoria "María Ferrer", Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Donación "Francisco Santojanni", Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Clínica Monte Grande, Monte Grande, Buenos Aires
  - Hospital Centro de Salud Zenón J. Santillán, San Miguel de Tucumán, Tucumán Province
  - Hospital San Juan de Dios, La Plata
- Spain (7):
  - Hospital de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

REFERENCES:
- [Derived] Agusti A, De Stefano G, Levi A, Munoz X, Romero-Mesones C, Sibila O, Lopez-Giraldo A, Plaza Moral V, Curto E, Echazarreta AL, Marquez SE, Pascual-Guardia S, Santos S, Marin A, Valdes L, Saldarini F, Salgado C, Casanovas G, Varea S, Rios J, Faner R. Add-on inhaled budesonide in the treatment of hospitalised patients with COVID-19: a randomised clinical trial. Eur Respir J. 2022 Mar 10;59(3):2103036. doi: 10.1183/13993003.03036-2021. Print 2022 Mar. PMID 35144989
- [Derived] Agusti A, Torres F, Faner R. Early treatment with inhaled budesonide to prevent clinical deterioration in patients with COVID-19. Lancet Respir Med. 2021 Jul;9(7):682-683. doi: 10.1016/S2213-2600(21)00171-5. Epub 2021 Apr 9. No abstract available. PMID 33844998
- [Derived] Farne H, Singanayagam A. Reply. J Allergy Clin Immunol. 2021 Mar;147(3):1117-1118. doi: 10.1016/j.jaci.2020.11.019. Epub 2020 Dec 30. No abstract available. PMID 33388170
- [Derived] Nicolau DV, Bafadhel M. Inhaled corticosteroids in virus pandemics: a treatment for COVID-19? Lancet Respir Med. 2020 Sep;8(9):846-847. doi: 10.1016/S2213-2600(20)30314-3. Epub 2020 Jul 30. No abstract available. PMID 32738928